CLINICAL TRIAL: NCT00775398
Title: A Phase 4, Multicenter, Open-Label, Observational Study Assessing the Impact of Exposure to THROMBIN-JMI® (Thrombin, Topical U.S.P [Bovine Origin]) on Coagulation Parameters
Brief Title: Observational Study Assessing the Impact of Exposure to THROMBIN-JMI® on Coagulation Parameters.
Acronym: MOSAIC
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: K847-08-4003
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Blood Coagulation
Keywords: Hemostasis; Thrombin-JMI; Thrombin; Blood Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: Subjects with anti-topical bovine thrombin antibodies pre-surgery, who received topical THROMBIN-JMI® during the study surgery.
- B: Subjects with anti-topical bovine thrombin antibodies pre-surgery, who did not received THROMBIN-JMI® during the study surgery.
- C: Subjects with no anti-topical bovine thrombin antibodies pre-surgery and who did receive THROMBIN-JMI® during the study surgery.
- D: Subjects with no anti-topical bovine thrombin antibodies pre-surgery and who did not receive THROMBIN-JMI® during the study surgery.

SUMMARY:
The purpose of this study is to assess the effect of possible exposure to THROMBIN JMI® on activated partial thromboplastin time (aPTT) at 48 hours post surgery in subjects with likelihood of prior exposure to THROMBIN JMI® within the past 4 years.

DETAILED DESCRIPTION:
This study is intended to observe the effects of possible repeat exposure to topical THROMBIN-JMI® on aPTT. Adult men and women who are scheduled to undergo qualified surgeries (defined as surgeries likely to require the use of an active topical hemostatic agent, but not likely to require transfusion of plasma), and who complete the informed consent process, and who meet all of the inclusion criteria and none of the exclusion criteria will be eligible for the study. As an observational study any decisions regarding the necessity for treatment to achieve hemostasis with this hemostatic product as an aid for perioperative hemostasis will be determined by the surgeon based upon the individual subject's condition.

Consequently, several assumptions and estimations are made in the design of the study. It is assumed that 20% of enrolled subjects will have pre-surgery bovine thrombin antibodies, and that 60% will receive THROMBIN JMI® during the study surgery, resulting in approximately 75 subjects in the primary study cohort and 195 subjects in the primary reference cohort. The primary endpoint of aPTT is chosen as prolongation beyond the normal reference range indicates either a factor deficiency or presence of an inhibitor. The latter is identified by either no correction or partial correction during mixing studies. At 48 hours post potential secondary exposure the secondary immune response should be sufficiently mounted as to see any impact of neutralizing antibodies on the aPTT.

After completion of the study surgeries, subjects will be categorized into cohorts based on whether their pre-surgery plasmas had or did not have anti-topical bovine thrombin antibodies and whether the subject received or did not receive THROMBIN JMI® intraoperatively. The primary study cohort will be subjects with anti-topical bovine thrombin antibodies pre-surgery, who received THROMBIN JMI® during the study surgery. The primary reference cohort will be those subjects with no anti-topical bovine thrombin antibodies pre-surgery and who did not receive THROMBIN JMI® during the study surgery. Antibody assessments will be not be performed until the end of the study for all subjects.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a subject MUST meet the following inclusion criteria:

* Must have undergone any one (or more) of the following surgical procedures within the past 4 years, but not less than 30 days before the study surgery: lumbar/cervical discectomy, lumbar/cervical laminectomy, microdiscectomy, shunt procedures, craniotomy, peripheral nerve surgical procedures, carotid artery surgery, repair of aneurysm, hip or other joint replacement, open repair of bone fracture, open spine procedures, creation of dialysis access, lower or upper extremity vascular bypass, skin grafting, burn wound debridement, facelift, abdominoplasty;
* Must be scheduled to undergo any one of the following surgical procedures, which is likely to require the use of topical thrombin, but is unlikely to require allogenic blood transfusion: lumbar/cervical discectomy, lumbar/cervical laminectomy, microdiscectomy, shunt procedures, craniotomy, peripheral nerve surgical procedures, carotid artery surgery, repair of aneurysm, hip or other joint replacement, open repair of bone fracture, open spine procedures, creation of dialysis access, lower or upper extremity revascularization, skin grafting, burn wound debridement, facelift, abdominoplasty;
* Must be 18 years of age or older;
* Must be capable and willing to provide written informed consent.

Exclusion Criteria:

To be eligible for this study, a subject MUST NOT meet any of the following exclusion criteria:

* Clinical history or clinical laboratory evidence of prior sensitivity to topical bovine thrombin, any of its components and/or other materials of bovine origin;
* A female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods and women who have been on hormonal contraceptives within 30 days of the surgical procedure;
* Medical condition or personal circumstances that will prevent participation in and completion of the follow-up visits at 48 hours, 4 weeks, and 8 weeks post-surgery;
* Currently participating in or has participated in (within 30 days prior to inclusion in this trial) another clinical trial of an investigational drug, biologic, device, or procedure;
* Known hematologic or medical condition that impedes/prolongs coagulation;
* Screening fibrinogen level less than the lower limit of normal based on the local laboratory ranges;
* Proposed exposure during the trial or previous known exposure to topical thrombin other than THROMBIN-JMI®;
* Prothrombin time, aPTT or TT outside of normal reference values at Baseline (e.g., Screening Visit).
* Planned use of therapeutic doses of intravenous heparin or low molecular weight heparin within 48 hours following surgery;
* Use of warfarin (Coumadin) within 5 days prior to surgery, or within 48 hours after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women who are scheduled to undergo qualified surgeries that are likely to require the use of an active topical hemostatic agent.
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in aPTT at 48 hours post surgery | Pre-surgery, 48 hours post-surgery

SECONDARY OUTCOMES:
Changes from Baseline in specified antibody levels at 48 hours, 4 weeks, and 8 weeks post-surgery | Pre-surgery, 48 hours, 4 weeks, 8 weeks post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Paterson, MD, MBA, Study Director — Medical Affairs
Locations (43):
- United States (43):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Arcadia, California
  - Glendale, California
  - Pasadena, California
  - San Diego, California
  - Boca Raton, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Muncie, Indiana
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Salisbury, Maryland
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Flint, Michigan
  - Grand Blanc, Michigan
  - Royal Oak, Michigan
  - Saginaw, Michigan
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Billings, Montana
  - Hackensack, New Jersey
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Sewickley, Pennsylvania
  - Fort Worth, Texas
  - Houston, Texas
  - Temple, Texas
  - Morgantown, West Virginia